CLINICAL TRIAL: NCT07326345
Title: Evaluation of the Effects of Different Rapid Maxillary Expansion Methods on the Nasomaxillary Complex Structures
Brief Title: Evaluation of Maxillary Expansion Methods on Nasomaxillary Structures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Merve Kulaksız (Other)
Responsible Party: Sponsor-Investigator, Merve Kulaksız, PhD student, Department of Orthodontics, Bezmialem Vakif University
Organization: Bezmialem Vakif University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E.211679
Record Dates: First submitted 2025-12-12; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Maxillary Expansion; Maxillary Transverse Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mini Screw-Supported Rapid Maxillary Expansion (MARPE) Group (Experimental)
  Interventions: Device: MARPE (Mini-Screw Assisted Rapid Palatal Expansion)
- Surgical-Assisted Rapid Maxillary Expansion (SARME) Group (Experimental)
  Interventions: Procedure: SARME (Surgically Assisted Rapid Maxillary Expansion)

INTERVENTIONS:
Device: MARPE (Mini-Screw Assisted Rapid Palatal Expansion) — A mini-screw assisted rapid palatal expansion device used to achieve skeletal maxillary expansion through bicortical anchorage. The device delivers orthopedic forces to the maxillary sutures with reduced dental tipping and greater skeletal effects compared to conventional rapid palatal expansion appliances.
  Arms: Mini Screw-Supported Rapid Maxillary Expansion (MARPE) Group
Procedure: SARME (Surgically Assisted Rapid Maxillary Expansion) — A surgically assisted maxillary expansion procedure performed to facilitate skeletal expansion in skeletally mature patients. The procedure involves weakening areas of resistance in the maxilla (e.g., lateral walls, midpalatal suture) followed by activation with a rapid palatal expansion device to achieve transverse maxillary widening.
  Arms: Surgical-Assisted Rapid Maxillary Expansion (SARME) Group

SUMMARY:
Maxillary transverse deficiency is an orthodontic anomaly characterized by the upper and lower dental arches being incompatible due to insufficient width of the maxilla. This condition typically manifests with clinical symptoms such as crossbite, crowding of teeth, and impaired respiratory function. Genetic factors, early primary tooth loss, mouth breathing, thumb sucking, and abnormal swallowing are among the causes of maxillary narrowing. Treatment options vary depending on the patient's age and the degree of suture closure. In pediatric and adolescent patients, rapid (RPE) or slow (SPE) orthodontic expansion can be achieved with palatal expansion appliances. However, in adult patients, due to the less flexible bone structure of the maxilla, methods such as surgically assisted expansion (SARME) or mini-screw-assisted expansion (MARPE) are preferred. Recent studies have shown that MARPE can be effective as a non-surgical alternative in young adults and can provide direct skeletal expansion without damaging the teeth.

DETAILED DESCRIPTION:
Thirty patients with maxillary transverse narrowing will be divided into two groups, MARPE and SARME, based on the amount of expansion required and suture ossification. Hybrid appliances will be custom-made for 15 patients undergoing mini-screw-supported rapid maxillary expansion. The position and number of screws will be determined individually for each patient. The screws to be used will have a diameter of 2 mm and a length of 14 mm. The screws will be placed under local anesthesia. A minimum of 2 and a maximum of 4 screws will be applied to patients. In the group undergoing surgical-assisted rapid maxillary expansion, expansion will be applied using an acrylic cap splint. In the SARME group, patients will undergo a standard Le Fort 1 osteotomy under general anesthesia. The appliances in both groups will be removed after a 6-month retention period. Cone beam computed tomography (90 kVp; 10 mA; 200 mm Voxel Size) will be taken from patients in both groups before starting the expansion treatment (T0) and after the 6-month retention period. Measurements will be performed on these radiological images using the Planmeca Romexis program. The volume, anteroposterior diameter, transverse diameter, length, and angle of the nasolacrimal canal and nasopalatine canal will be measured before and after treatment. The volume of the maxillary sinus and the diameter of the ostium openings will be measured. The nasal breathing volume and septal deviation will be measured on CBCT before treatment (T0) and at the end of the retention period (T1), and the results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of maxillary transverse deficiency.
* Patients aged 15 years and older.
* Presence of unilateral or bilateral crossbite.

Exclusion Criteria:

* Severe facial deformities or craniofacial syndromes.
* History of previous orthodontic treatment.
* Existing pathology or history of surgery related to the paranasal sinuses, nasolacrimal system, or orbital cavity.
* Inadequate patient cooperation.
* History of trauma, or previous maxillofacial/plastic surgery procedures.
* Clinical signs or symptoms of maxillary sinus pathology (e.g., maxillary sinus cysts, sinusitis).

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Changes in Craniofacial Volumes | Cone-beam computed tomography (CBCT) scans will be obtained from patients in both groups at two specific time points: before the initiation of expansion treatment (T0) and following the 6-month retention period (T1).
  Evaluation of volumetric changes using CBCT analysis. Specific measurements include the total volume of the nasolacrimal and nasopalatine canals, maxillary sinus volume, and nasal airway volume.
Changes in Linear Dimensions of Canals and Ostium | Before expansion (T0) and after 6-month retention (T1).
  Assessment of linear changes including the anteroposterior and transverse diameters and lengths of the nasolacrimal and nasopalatine canals. Additionally, the diameter of the maxillary sinus ostium openings will be measured in millimeters.
Changes in Angulation and Septal Deviation | Cone-beam computed tomography (CBCT) scans will be obtained from patients in both groups at two specific time points: before the initiation of expansion treatment (T0) and following the 6-month retention period (T1).
  Assessment of angular changes in craniofacial structures. This includes the angulation of the nasolacrimal and nasopalatine canals and the degree of nasal septal deviation.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University Faculty of Dentistry, Department of Orthodontics, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No